CLINICAL TRIAL: NCT00370318
Title: Multicentre Study to Assess the Effect of Prophylactic Antipyretic Treatment on the Rate of Febrile Reactions Following Concomitant Administration of GSK Biologicals' 10-valent Pneumococcal Conjugate, Infanrix Hexa and Rotarix Vaccines
Brief Title: Prophylactic Antipyretic Treatment in Children Receiving Pneumococcal Conjugate and Standard Infant Vaccines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 107017
Record Dates: First submitted 2006-06-02; First posted 2006-08-31 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Infections, Rotavirus
Keywords: Pneumococcal Disease
MeSH Terms: conditions — Rotavirus Infections; Pneumococcal Infections | interventions — 10-valent pneumococcal conjugate vaccine; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; RIX4414 vaccine; Acetaminophen

INTERVENTIONS:
Biological: 10 valent pneumococcal conjugate vaccine
Biological: Infanrix Hexa
Biological: Rotarix
Drug: Paracetamol
  Other Names: Rotarix; Infanrix Hexa; 10 valent pneumococcal conjugate vaccine

SUMMARY:
The purpose of this trial is to assess if the rate of febrile reactions following the co-administration of pneumococcal conjugate vaccines with standard infant vaccines is lowered when paracetamol is given prophylactically.

DETAILED DESCRIPTION:
2 groups (200 per group); control group receives no prophylactic antipyretic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children 9-16 weeks old and born after a gestation of at least 36 weeks.

Exclusion Criteria:

* Body weight < 4.5 kg
* Children having received or planning to receive any investigational or non-registered products, vaccines not foreseen in the protocol, and immune modifying drugs
* Children with any disease that affects the immune system or gastro-intestinal tract
* Children with a history of seizures, allergic disease, or disease(s) covered by the vaccines
* Children with contraindication to paracetamol treatment.

Ages: 9 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400
Dates: Start 2006-09; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of fever > or = to 38°C (rectal temperature)

SECONDARY OUTCOMES:
Safety, reactogenicity and immunogenicity pre and post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Czechia (8):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Jindřichův Hradec
  - GSK Investigational Site, Náchod
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Znojmo

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Prymula R, Siegrist CA, Chlibek R, Zemlickova H, Vackova M, Smetana J, Lommel P, Kaliskova E, Borys D, Schuerman L. Effect of prophylactic paracetamol administration at time of vaccination on febrile reactions and antibody responses in children: two open-label, randomised controlled trials. Lancet. 2009 Oct 17;374(9698):1339-50. doi: 10.1016/S0140-6736(09)61208-3. PMID 19837254
- [Background] Schuerman L, Borys D, Hoet B, Forsgren A, Prymula R. Prevention of otitis media: now a reality? Vaccine. 2009 Sep 25;27(42):5748-54. doi: 10.1016/j.vaccine.2009.07.070. Epub 2009 Aug 8. PMID 19666154
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 107017 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107017 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 107017 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107017 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 107017 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107017 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register